CLINICAL TRIAL: NCT01171014
Title: A Three-Arm, Placebo Controlled, Double-Blind, Single Center Study to Evaluate the Impact of Probiotic Strain Bifidobacterium Lactis HN019 on Intestinal Well-Being, Colonic Transit Time and Digestive Discomfort
Brief Title: Effect of Bifidobacterium Lactis HN019 on Colonic Transit Time and Digestive Symptoms
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Fonterra Research Centre (Industry)
Collaborators: Danisco (Industry); Sprim Advanced Life Sciences (Other)
Responsible Party: Pramod Gopal，PhD, Fonterra Research Centre
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: #08-SPUS-o6-FON-01
Record Dates: First submitted 2010-07-26; First posted 2010-07-28 (Estimated); Last update posted 2010-07-28 (Estimated); Status verified 2010-07

CONDITIONS: Gastrointestinal Symptoms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- High dose probiotic (Experimental): Bifidobacterium lactis HN019, 10 billion cfu/day
  Interventions: Dietary Supplement: Bifidobacterium lactis HN019
- Low dose probiotic (Experimental): Bifidobacterium lactis HN019, 1 billion cfu/day
  Interventions: Dietary Supplement: Bifidobacterium lactis HN019
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Bifidobacterium lactis HN019 — Bifidobacterium lactis HN019, 10 billion cfu/day, once a day for 14 days
  Arms: High dose probiotic
Dietary Supplement: Bifidobacterium lactis HN019 — Bifidobacterium lactis HN019, 1 billion cfu/day, once a day for 14 days
  Arms: Low dose probiotic
Dietary Supplement: Placebo — Placebo, once a day for 14 days
  Arms: Placebo

SUMMARY:
The purpose of this study was to investigate the dose response effect of Bifidobacterium lactis HN019 supplementation on colonic transit time and gastrointestinal symptoms.

ELIGIBILITY:
Inclusion Criteria:

* healthy males and females aged 25 to 65 years
* stool type 2-4 on the Bristol Stool Chart
* 1 to 3 bowel movements per week

Exclusion Criteria:

* use of any probiotic product intended to improve gastrointestinal function within the 2 weeks preceding study entry
* major chronic and uncontrolled systemic medical conditions
* severe gastrointestinal conditions known to prolong CTT
* lactose intolerance
* chronic diarrhea
* gastric bypass surgery or lap band insertion for weight loss
* regular laxative use
* pregnant or breast-feeding women

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2009-06; Primary Completion 2009-12 (Actual); Study Completion 2009-12 (Actual)

PRIMARY OUTCOMES:
Colonic transit time | 14 days

SECONDARY OUTCOMES:
Gastrointestinal symptoms | 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Philip Waller, MD, Principal Investigator — Accurate Clinical Research, Houston, TX